CLINICAL TRIAL: NCT00004210
Title: Outcomes in Education and Counseling for HNPCC Testing
Brief Title: Study of the Results of Education and Counseling for Persons Undergoing Genetic Testing for Hereditary Nonpolyposis Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDR0000067459; NCI-95-HG-0165; NCI-NMOB-9501; NHGRI-95-HG-0165; NCT00001470 (obsolete NCT alias)
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling

INTERVENTIONS:
Other: loss of heterozygosity analysis
Other: microsatellite instability analysis
Other: mutation analysis
Other: counseling intervention

SUMMARY:
RATIONALE: Identifying family and individual characteristics may help plan education and counseling for patients who are considering genetic testing.

PURPOSE: This clinical trial is studying education and counseling to see what effect they have in patients who are undergoing genetic testing for hereditary nonpolyposis colon cancer (recruitment of new families with HNPCC stopped as of 04-26-06, recruitment of persons within families already participating continues).

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify family characteristics, personality traits, and religious and spiritual beliefs that significantly affect individual decisions regarding mutation testing for hereditary nonpolyposis colon cancer (HNPCC) (recruitment of new families with HNPCC stopped as of 04-26-06, recruitment of persons within families already participating continues).
* Determine the impact of negative vs positive mutation test results on family relationships and psychological status.
* Assess expectations regarding testing and how they influence perceptions of risks and responses to risk notification.
* Determine the impact of risk notification on the frequency of screening/prevention activities.
* Formulate a standard diagnostic algorithm for determining microsatellite instability based on the analysis of tumors with this extensive array of markers and correlate specific replication error phenotypes with germline genotype.

OUTLINE: Participants complete a baseline assessment of knowledge, risk perception, and personality traits followed by a structured pretest education session. Participants are then offered the choice of whether or not to undergo genetic testing for mutations in hereditary nonpolyposis colon cancer (HNPCC) genes. Participants who choose to undergo genetic testing provide a blood sample for this purpose. Participants who undergo genetic testing receive results and counseling (recruitment of new families with HNPCC stopped as of 04-26-06, recruitment of persons within families already participating continues).

Available surveillance options are discussed for all participants. Psychological and behavioral outcomes are reassessed at 6 and 12 months for both those choosing and not choosing genetic testing.

Tumors (when available) are analyzed for mismatched repair deficiency on the basis of microsatellite instability.

PROJECTED ACCRUAL: A total of 900 participants will be accrued for this study, with a specific target of 200 individuals who have not experienced cancer within families identified with hereditary nonpolyposis colon cancer (HNPCC) mutations (recruitment of new families with HNPCC stopped as of 04-26-06, recruitment of persons within families already participating continues).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Family history consistent with hereditary nonpolyposis colon cancer (HNPCC)*

    * At least 3 relatives with histologically proven colorectal cancer or HNPCC-associated cancer and 1 is a first-degree relative of the other 2
    * At least 2 successive generations affected
    * Colorectal cancer (or HNPCC-associated cancer) diagnosed under age 50 in 1 of the relatives
  * Diagnosis of colorectal cancer under age 41
  * HNPCC-associated cancer/polyps* under age 41 with a microsatellite instability (MSI) phenotype
  * Multiple primary HNPCC-associated cancers* regardless of family history
  * Colorectal or other HNPCC-associated tumor/polyp* demonstrating a positive MSI phenotype and at least 1 second-degree (or closer) and 1 third-degree (or closer) relative with a HNPCC-associated cancer

    * 1 affected family member must have one of the following:

      * Right-sided colon cancer
      * Multiple primary HNPCC-associated cancers
      * Diagnosis of cancer prior to age 51 NOTE: *Recruitment of new families with HNPCC stopped as of 04-26-06, recruitment of persons within families already participating continues

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2000-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Assessment of cancer risk perception, cancer screening practices, views regarding genetic services, and family communication about HNPCC / Lynch syndrome by family members

CONTACTS AND LOCATIONS:
Overall Officials: Donald W. Hadley, MS, CGC, Study Chair — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - National Human Genome Research Institute, Bethesda, Maryland

REFERENCES:
- [Result] Hadley DW, Ashida S, Jenkins JF, Calzone KA, Kirsch IR, Koehly LM. Colonoscopy use following mutation detection in Lynch syndrome: exploring a role for cancer screening in adaptation. Clin Genet. 2011 Apr;79(4):321-8. doi: 10.1111/j.1399-0004.2010.01622.x. Epub 2011 Jan 19. PMID 21204803
- [Result] Hadley DW, Jenkins JF, Dimond E, de Carvalho M, Kirsch I, Palmer CG. Colon cancer screening practices after genetic counseling and testing for hereditary nonpolyposis colorectal cancer. J Clin Oncol. 2004 Jan 1;22(1):39-44. doi: 10.1200/JCO.2004.06.128. PMID 14701766
- [Result] Hadley DW, Jenkins J, Dimond E, Nakahara K, Grogan L, Liewehr DJ, Steinberg SM, Kirsch I. Genetic counseling and testing in families with hereditary nonpolyposis colorectal cancer. Arch Intern Med. 2003 Mar 10;163(5):573-82. doi: 10.1001/archinte.163.5.573. PMID 12622604
- [Derived] Hadley DW, Eliezer D, Addissie Y, Goergen A, Ashida S, Koehly L. Uptake and predictors of colonoscopy use in family members not participating in cascade genetic testing for Lynch syndrome. Sci Rep. 2020 Sep 29;10(1):15959. doi: 10.1038/s41598-020-72938-z. PMID 32994442